CLINICAL TRIAL: NCT03246373
Title: Prospective, Single Center, Observational, Clinical Trial of the Effects of Cerebral Collateral Circulation on the Outcome of Leukoaraiosis in High-risk Population
Brief Title: the Effects of Cerebral Collateral Circulation on the Outcome of Leukoaraiosis in High-risk Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSA2016KY001
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Leukoaraiosis
Keywords: cognitive impairment
MeSH Terms: conditions — Leukoaraiosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood sample fingernail sample hair sample urinary sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study observed the relationship between cerebral collateral circulation and the prognosis of leukoaraiosis in high-risk population. Cerebral collateral circulation and leukoaraiosis levels will be evaluated and followed up by magnetic resonance examination. The participants' clinical performance caused by leukoaraiosis will be assessed by a series of scales.

DETAILED DESCRIPTION:
1. Case collection information is sent daily to clinical trial supervisors.
2. The clinical trial team meets once a week to monitor the quality of clinical trials.
3. The severity of the leukoaraiosis will be evaluated by a scale. The patients whose score is more than 2 will take additional magnetic resonance examination including magnetic resonance angiography (MRA) and arterial spin labeling (ASL). And their cognitive ability will be evaluated by a series of scales including Mini-Mental State Examination (MMSE) and Montreal cognitive assessment (MoCA) and gait by the short physical performance battery (SPPB).

   The blood sample will be taken for biochemical detection and hair and nail samples for trace element detection.
4. Data were analyzed by regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Physical Examinees or out-patients
* The MRI scale score ≥ 2

Exclusion Criteria:

* History of stroke
* History of malignant tumor
* History of connective tissue disease
* Pregnant, trying to become pregnant or within 6 weeks after delivery
* serious infections

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients of physical exmination department or out-patients of neurology department in Zhongshan hospital Fudan University.
Sampling Method: Probability Sample
Enrollment: 1037 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
change in cognitive assessment scale score | baseline and one year
  It will be assessed by the Mini-Mental state examination (MMSE) and Montreal cognitive assessment (MoCA). Each assessment is scored 0-30, yielding a total between 0-60.

SECONDARY OUTCOMES:
change in mood assessment Scale score | baseline and one year
  It will be assessed by Hamilton Depression Scale (HAMD). It is scored 0-30.
change in gait evaluation score | baseline and one year
  It will be assessed by the short physical performance battery (SPPB). It is scored 0-11.
stroke | baseline and one year
  The participant is diagnosed with stroke

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — neurology department of Zhongshan hospital, Fudan University
Locations (1):
- neurology department of Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No